CLINICAL TRIAL: NCT04841824
Title: Dysfunction and Endothelial Repair in Sepsis Shock : RNAseq Transcriptomic Analysis of Circulating Endothelial Cells
Brief Title: TRanscriptomic Analysis of Circulating Endothelial Cells During Sepsis - TRACES Study
Acronym: TRACES
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201060
Record Dates: First submitted 2021-04-02; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Critical Illness With or Without Sepsis
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Critically ill patients with sepsis
  Interventions: Other: Observational study
- Critically ill patients without sepsis

INTERVENTIONS:
Other: Observational study — Observational study. Groups are defined based on baseline patients' characteristics : presence or absence of sepsis.
  Groups: Critically ill patients with sepsis

SUMMARY:
Vascular dysfunction is an important mechanism involved in organ failure, in the setting of sepsis condition, with different types of circulating endothelial cells.Transcriptom analysis via RNAseq in different types of circulating endothelial cells, comapring critically ill patients with or without sepsis will allow determining differential gene expression for signal pathways in endothelial alteration and restoration associated with sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years
* Admission in intensive care with or without sepsis
* Health insurance as per the national insurance system
* Informed and unopposed patient for participation (or referend closed one)

Exclusion Criteria:

* Patient under legal protection
* Patient under national medical help system
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adult patients hospitalized in an intensive care unit, with or without sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Gene expression based on transcriptom analysis of circulating endothelial cells | Day 1
  Gene expression based on transcriptom analysis of circulating endothelial cells (RNAseq)

SECONDARY OUTCOMES:
Counts of circulating endothelial cells | Day 1 and Day 3
  Counts of circulating endothelial cells, including progenitor cells
Sequential Organ Failure Assessment (SOFA) score | Day 1, Day 3, Day 7
  Sequential Organ Failure Assessment (SOFA) score, ranging from 0 (best: absence of organ failure) to 24 (worse: multiple organ failure)
Sequential Organ Failure Assessment (SOFA) hemodynamic sub-score | Day 1, Day 3, Day 7
  Sequential Organ Failure Assessment (SOFA) hemodynamic sub-score, ranging from 0 (best: absence of hemodynamic failure) to 4 (worse: hemodynamic failure)
Sequential Organ Failure Assessment (SOFA) respiratory sub-score | Day 1, Day 3, Day 7
  Sequential Organ Failure Assessment (SOFA) respiratory sub-score, ranging from 0 (best: absence of respiratory failure) to 4 (worse: respiratory failure)
Sequential Organ Failure Assessment (SOFA) neurological sub-score | Day 1, Day 3, Day 7
  Sequential Organ Failure Assessment (SOFA) neurological sub-score, ranging from 0 (best: absence of neurological failure) to 4 (worse: neurological failure)
Sequential Organ Failure Assessment (SOFA) hematological sub-score | Day 1, Day 3, Day 7
  Sequential Organ Failure Assessment (SOFA) hematological sub-score, ranging from 0 (best: absence of hematological failure) to 4 (worse: hematological failure)
Intensive care unit (ICU) mortality | ICU length of stay
  Death during ICU stay
D28 mortality | Day 28
  Death within 28 days of intensive care unit
Hospital mortality | Day 90
  Death within 90 days of intensive care unit
Duration of ventilation | Day 28
  Number of days alive without ventilation up to Day 28
Duration of renal replacement therapy (RRT) | Day 28
  Number of days alive without RRT up to Day 28
Duration of vasopressors therapy | Day 28
  Number of days alive without vasopressors up to Day 28
Dose of vasopressors | ICU length of stay, assessed up to 90 days
  Dose of vasopressors, in patients who received vasopressors
Duration of intensive care unit (ICU) stay | Day 28
  Number of days alive outside the ICU up to D28
Circulating endothelial cells cytokines profile | Day 1 and 3
  Dosage of cytokines from circulating endothelial cells
Circulating endothelial cells chemokines profile | Day 1 and 3
  Dosage of chemokines from circulating endothelial cells
Expression of membrane proteins of endothelial cells | Day 1 and 3
  Expression of membrane proteins of endothelial cells by flow cytometry
Infection site | Day 1
  Infection site for patients with sepsis
Infection identification | Day 1
  Identified germs for patients with sepsis
Number of participants with different types of antibiotic treatment | Length of ICU stay, assessed up to 90 days
  Antibiotic treatments for patients with sepsis during intensive care unit (ICU) stay

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP Hôpital Saint Louis, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided